CLINICAL TRIAL: NCT04103736
Title: The Effect of Dietary Nitrates on Physical Performance and Vascular Function in Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 706281-6
Record Dates: First submitted 2019-04-29; First posted 2019-09-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Kidney Disease, Chronic; Endothelial Dysfunction
Keywords: chronic kidney disease; dietary nitrates; beetroot juice; endothelium, vascular; cardiovascular disease; exercise capacity
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beet Juice Supplement (Experimental): A single, acute dose of Beet It Sport Shot containing ~12.6mmol naturally occurring dietary nitrates.
  Interventions: Dietary Supplement: Beet It Sport Shot
- Placebo juice (Placebo Comparator): A single, acute dose of nitrate-depleted Beet It Sport Shot
  Interventions: Dietary Supplement: Nitrate-depleted placebo

INTERVENTIONS:
Dietary Supplement: Beet It Sport Shot — Source of naturally occurring dietary nitrates
  Arms: Beet Juice Supplement
Dietary Supplement: Nitrate-depleted placebo — Placebo
  Arms: Placebo juice

SUMMARY:
The purpose of this study is to examine the effect of acute ingestion of a concentrated beetroot juice supplement on vascular function and exercise capacity in patients with moderate to severe chronic kidney disease

DETAILED DESCRIPTION:
People with Chronic Kidney Disease (CKD) are at an increased risk of cardiovascular disease. Blood vessel dysfunction and exercise intolerance are common in CKD. Blood vessel dysfunction has been shown to predict future cardiovascular events and decreased physical activity can contribute to an increased risk of cardiovascular disease. Therefore, this study investigates if dietary nitrate from beetroot juice, which has been shown to improve blood vessel function and exercise capacity in other cardiovascular disease pathologies, could be effective at improving these measures in patients with CKD. In a controlled, double blinded trial, stage 3-5 CKD patients will be randomly assigned to receive either beetroot beverage or a placebo and then complete measures of blood vessel function and an exercise test.

ELIGIBILITY:
Inclusion Criteria:

• Stage 3-5 Chronic Kidney Disease

Exclusion Criteria:

* History of cardiovascular disease
* Current pregnancy
* Uncontrolled hypertension
* Uncontrolled hyperlipidemia
* Current hormone replacement therapy
* Current use of tobacco products
* Current autoimmune disease
* Current hyperkalemia
* Diagnosis of a deep vein thrombosis (DVT) within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2017-06-29 (Actual); Study Completion 2017-06-29 (Actual)

PRIMARY OUTCOMES:
Microvascular Function, assessed by laser Doppler flowmetry coupled with intradermal microdialysis | 2.5 hours post ingestion of juice
  Nitric oxide mediated cutaneous microvascular dilatory response to local heating assessed by laser Doppler flowmetry coupled with microdialysis

SECONDARY OUTCOMES:
Endothelial function | 2.5 hours post ingestion of juice
  Conduit artery endothelial function assessed by brachial artery flow mediated dilation
Blood pressure | Change from pre-ingestion baseline to 2.5 hours post ingestion of juice
  Blood pressure recorded by automatic blood pressure machine
Arterial stiffness | 2.5 hours post ingestion of juice
  Carotid to femoral pulse wave velocity assessed by tonometry
Pulse wave analysis | 2.5 hours post ingestion of juice
  Central blood pressure and augmentation index assessed by oscillometry and radial tonometry
Peak aerobic capacity | 2.5 hours post ingestion of juice
  Peak oxygen uptake (VO2 peak) during incremental cycling exercise to exhaustion

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Kinesiology and Applied Physiology, University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No